## **Cover Page for Statistical Analysis Plan**

| Sponsor-Investigator: | Barry London |
|-----------------------|------------------------------------|
| NCT Number: | NCT02441101 |
| Unique Protocol ID: | 201409760 |
| Official Title: | Right Ventricular Septal Pacing in |
| | Patients With Right Bundle Branch |
| | Block and Heart Failure (The |
| | SPARK Trial) |
| Date of Document: | 24 December 2014 |

Linear mixed model analysis for repeated measures will be used to test for change over the follow-up period in the primary outcome measures. Post-hoc pairwise comparison with baseline will be performed using Dunnett's test. Mean estimates at each time point, and mean change from baseline (with 95% confidence limits) will be computed from the fitted model. All tests were two-tailed and a p < 0.05 was considered as statistically significant. All analyses will be conducted using the intention-to-treat population.